CLINICAL TRIAL: NCT06067854
Title: Perioperative Analgesia in Neonates Who Underwent Primary Cleft Lip Repair Surgery: Retrospective Study
Brief Title: Perioperative Analgesia in Neonates Who Underwent Primary Cleft Lip Repair Surgery
Status: Completed | Type: Observational
Sponsor: Brno University Hospital (Other)
Collaborators: Masaryk University (Other)
Responsible Party: Principal Investigator, Petr Štourač, MD, Clinical Professor, Brno University Hospital
Other Study IDs: KDAR 9/2023
Record Dates: First submitted 2023-09-28; First posted 2023-10-05 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Perioperative Analgesia in Neonates
Keywords: perioperative analgesia; primary cleft lip repair surgery; infraorbital peripheral blockade
MeSH Terms: interventions — Anesthesia, Conduction; Surgeons

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Neonates under general anaesthesia without regional anaesthesia: the standard procedure - without regional anaesthesia
- Neonates under general anaesthesia with regional anaesthesia: infraorbital peripheral blockade with or without nasal peripheral blockade according to the preference of the anesthesiologist and surgeon

INTERVENTIONS:
Procedure: the standard procedure - without regional anaesthesia — the standard procedure - without regional anaesthesia
Procedure: infraorbital peripheral blockade with or without nasal peripheral blockade according to the preference of the anesthesiologist and surgeon — infraorbital peripheral blockade with or without nasal peripheral blockade according to the preference of the anesthesiologist and surgeon

SUMMARY:
In retrospective data search the investigators will identified the cumulative consumption of opioid analgesics during surgery and 24 hours after surgery in neonate with cleft lips who underwent primary cleft lip repair surgery.

DETAILED DESCRIPTION:
The cumulative consumption of opioids during surgery and 24 hours after surgery in neonates with cleft lips who underwent primary cleft lip repair surgery is not known. Patients were divided into two groups according to the time period when they underwent surgery. Group 1 were neonates who underwent primary cleft lip repair surgery under general anaesthesia without regional anaesthesia - the time period before regional anesthesia is introduced into the standard procedure. Group 2 are newborns who underwent primary cleft lip repair surgery under general anaesthesia with regional anaesthesia. Group 1 underwent surgery in time period before regional anesthesia was introduced into the standard procedure. In this retrospective study, the anesthesiology perioperative data from January 2018 till December 2021 in the tertiary center of Pediatric anaesthesia will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* neonates with unilateral or bilateral cleft lip (U/BCL), all neonates with unilateral or bilateral cleft lip and alveolus (U/BCLA) or with unilateral or bilateral cleft lip, alveolus and palate (total cleft; U/BCLAP) who underwent cleft lip repair surgery in the neonatal period
* the study period (1/2018-12/2021)

Exclusion Criteria:

* ● presence of coagulopathy

  * thrombocytopenia or thrombopathy
  * patients at risk of malignant hyperthermia
  * patients who were not neonates (older than 28 days)
  * patients who required postoperative mechanical ventilation

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates with cleft lips who underwent primary cleft lip repair surgery in tertiary center paediatric anesthesiology department
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
The cumulative consumption of opioids during surgery and 24 hours after surgery | 24 hours after surgery
  The cumulative consumption of opioid analgesics during surgery and 24 hours after surgery in neonates with regional block compared to neonates without regional anesthesia

SECONDARY OUTCOMES:
Oral intake | 24 hours after surgery
  Difference in time of first oral intake after surgery in the group with regional anesthesia compared to with the group without regional anaesthesia
Complications | 24 hours after surgery
  Complications of regional anesthesia including suction disorders in the group with regional anaesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Petr Stourac, prof. MD., Ph.D., MBA, Study Chair — Department of paediatric anaesthesia and intensive care medicine
Locations (1):
- Brno University Hospital, Brno, South Moravian, Czechia

REFERENCES:
- [Derived] Richtrova M, Koskova O, Janku M, Bonischova T, Fabian D, Stourac P. Regional anesthesia in neonates with cleft lip and palate: Retrospective study. Int J Pediatr Otorhinolaryngol. 2024 May;180:111965. doi: 10.1016/j.ijporl.2024.111965. Epub 2024 May 4. PMID 38718430